CLINICAL TRIAL: NCT00639678
Title: A Randomized, Single-blind, Placebo-controlled Study to Evaluate the Safety and Tolerability of Raxibacumab (Human Monoclonal Antibody to B. Anthracis Protective Antigen) in Healthy Subjects
Brief Title: A Study to Evaluate the Safety and Tolerability of Raxibacumab in Healthy Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Human Genome Sciences Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry); Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HGS1021-C1063; NCT02075814 (obsolete NCT alias)
Record Dates: First submitted 2008-03-13; First posted 2008-03-20 (Estimated); Results first posted 2014-02-07 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2014-01

CONDITIONS: Healthy
Keywords: healthy volunteers
MeSH Terms: interventions — raxibacumab

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: raxibacumab
- 2 (Experimental)
  Interventions: Drug: raxibacumab
- 3 (Placebo Comparator)
  Interventions: Drug: placebo
- 4 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — 40 mg/kg intravenously, double dose (day 0 and 14), Group 3
  Arms: 3
Drug: raxibacumab — 40 mg/kg intravenously, double dose (day 0 and 14), Group 1
  Arms: 1
Drug: placebo — 40 mg/kg placebo, single dose (day 0), Group 4
  Arms: 4
Drug: raxibacumab — 40 mg/kg intravenously, single dose, day 0, Group 2
  Arms: 2

SUMMARY:
To evaluate the safety and tolerability of raxibacumab in healthy subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, 18 years of age or older
* Normal laboratory (blood test) results
* Subjects are eligible to enter the study if they are not pregnant or nursing, are sterile or of non-childbearing potential, or are willing to practice abstinence or use appropriate birth control methods during the study (about 2 months)

Key Exclusion Criteria:

* History of significant, acute or chronic diseases (ie, heart, lung, gastrointestinal, liver, kidney, neurological or infectious diseases).
* Prior immunization with anthrax vaccine adsorbed (AVA), prior treatment with investigational anthrax therapies, prior treatment for anthrax exposure, or prior anthrax infection.
* History of Type I hypersensitivity reaction to food or drugs, IV contrast agents, antihistamines, or history of hives.
* A current drug or alcohol addiction.
* Positive for human immunodeficiency virus (HIV-1), Hepatitis B surface antigen, or Hepatitis C antibody.
* Cancer within the last 5 years (with the exception of adequately treated basal cell carcinoma of the skin or in situ carcinoma of the cervix).
* Participation within 60 days of intiating study or refusal to refrain from participation during the study in any other clinical trials of an investigational compound.
* Previous exposure to raxibacumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2008-03; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Migone TS, Subramanian GM, Zhong J, Healey LM, Corey A, Devalaraja M, Lo L, Ullrich S, Zimmerman J, Chen A, Lewis M, Meister G, Gillum K, Sanford D, Mott J, Bolmer SD. Raxibacumab for the treatment of inhalational anthrax. N Engl J Med. 2009 Jul 9;361(2):135-44. doi: 10.1056/NEJMoa0810603. PMID 19587338

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized to a treatment group at a ratio of 3:1 (raxibacumab:placebo). Participants were randomized to the double dose cohorts first. When randomization was completed for the double-dose cohorts, participants were then randomized into the single-dose cohorts.
Pre-assignment Details: A total of 322 participants were randomized and 320 participants were administered at least one dose of study treatment.
Groups:
- Placebo - Single-Dose: Participants received a single dose of placebo administered via intravenous (IV) infusion. Participants were treated with oral diphenhydramine (25-50 milligrams [mg]) up to 60 minutes prior to infusion of placebo.
- Placebo - Double-Dose: Participants received a double dose of placebo administered 14 days apart via IV infusion. Participants were treated with oral diphenhydramine (25-50 mg) up to 60 minutes prior to infusion of placebo.
- Raxibacumab - Single-Dose: Participants received a single dose of 40 mg/kilogram (kg) raxibacumab administered via IV infusion. Participants were treated with oral diphenhydramine (25-50 mg) up to 60 minutes prior to infusion of raxibacumab.
- Raxibacumab - Double-Dose: Participants received a double dose of 40 mg/kg raxibacumab administered 14 days apart via IV infusion. Participants were treated with oral diphenhydramine (25-50 mg) up to 60 minutes prior to infusion of raxibacumab.
Period: Overall Study
Arm/Group | Placebo - Single-Dose | Placebo - Double-Dose | Raxibacumab - Single-Dose | Raxibacumab - Double-Dose
Started | 74 | 6 | 217 | 23
Completed | 70 | 5 | 206 | 23
Not Completed | 4 | 1 | 11 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 4 | 0
Not completed — Lost to Follow-up | 1 | 0 | 6 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Lack of Compliance | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo - Single-Dose | Placebo - Double-Dose | Raxibacumab - Single-Dose | Raxibacumab - Double-Dose | Total
Number analyzed (Participants) | 74 | 6 | 217 | 23 | 320
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.8 (16.8) | 52.2 (13.8) | 40.3 (16.3) | 48.5 (14.6) | 41.0 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 4 | 117 | 13 | 164
  Male | 44 | 2 | 100 | 10 | 156
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 57 | 4 | 143 | 21 | 225
  Asian | 4 | 0 | 15 | 0 | 19
  Black or African American | 4 | 2 | 21 | 1 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 0 | 2
  Not Listed | 0 | 0 | 1 | 0 | 1
  Multiracial | 2 | 0 | 7 | 0 | 9
  Hispanic or Latino origin | 7 | 0 | 28 | 1 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) or Any Serious Adverse Event (SAE) During the Treatment Period
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. This includes worsening (eg, increase in frequency or severity) of pre-existing conditions. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. Medical or scientific judgment should be exercised in deciding whether reporting is appropriate in other situations. Refer to the General Adverse AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From the day of the first dose of study agent (Day 0) until Day 56 (single-dose) or until Day 70 (double-dose)
Population: As-treated population: all participants who received at least one dose of study agent, with the assignment to treatment based on the actual treatment received, unless otherwise specified
Measure: Number; unit: Participants
Groups:
- Raxibacumab - Single-Dose: Participants received a single dose of 40 milligrams (mg)/kilogram (kg) raxibacumab administered via IV infusion. Participants were treated with oral diphenhydramine (25-50 mg) up to 60 minutes prior to infusion of raxibacumab.
Arm/Group | Placebo - Single-Dose | Placebo - Double-Dose | Raxibacumab - Single-Dose | Raxibacumab - Double-Dose
Number analyzed (Participants) | 74 | 6 | 217 | 23
Participants
  Any AE | 32 | 6 | 103 | 10
  Any SAE | 0 | 1 | 0 | 1

2. Primary Outcome: Number of Participants With Hematological Toxicities of the Indicated Grade
Description: Clinical hematological parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable.
Time Frame: From the day of the first dose of study agent (Day 0) until Day 56 (single-dose) or until Day 70 (double-dose)
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Placebo - Single-Dose | Placebo - Double-Dose | Raxibacumab - Single-Dose | Raxibacumab - Double-Dose
Number analyzed (Participants) | 74 | 6 | 217 | 23
Participants
  Leukocytosis, Grade 1 | 4 | 0 | 15 | 2
  Leukocytosis, Grade 2 | 1 | 0 | 2 | 2
  Leukocytosis, Grade 3 | 1 | 0 | 1 | 0
  Leukocytosis, Grade 4 | 0 | 0 | 0 | 0
  Leukopenia, Grade 1 | 9 | 1 | 25 | 4
  Leukopenia, Grade 2 | 1 | 0 | 6 | 0
  Leukopenia, Grade 3 | 0 | 0 | 0 | 0
  Leukopenia, Grade 4 | 0 | 0 | 0 | 0
  Neutropenia, Grade 1 | 4 | 0 | 8 | 1
  Neutropenia, Grade 2 | 1 | 0 | 1 | 0
  Neutropenia, Grade 3 | 0 | 0 | 0 | 0
  Neutropenia, Grade 4 | 0 | 0 | 1 | 0
  Lymphopenia, Grade 1 | 1 | 0 | 3 | 0
  Lymphopenia, Grade 2 | 0 | 0 | 1 | 0
  Lymphopenia, Grade 3 | 0 | 0 | 0 | 0
  Lymphopenia, Grade 4 | 0 | 0 | 0 | 0
  Hemoglobin, Grade 1 | 1 | 0 | 12 | 0
  Hemoglobin, Grade 2 | 0 | 0 | 0 | 0
  Hemoglobin, Grade 3 | 0 | 0 | 0 | 0
  Hemoglobin, Grade 4 | 0 | 0 | 0 | 0
  Platelet, Grade 1 | 0 | 0 | 0 | 0
  Platelet, Grade 2 | 0 | 0 | 0 | 0
  Platelet, Grade 3 | 0 | 0 | 0 | 0
  Platelet, Grade 4 | 0 | 0 | 0 | 0
  Prothrombin Time, Grade 1 | 0 | 0 | 2 | 0
  Prothrombin Time, Grade 2 | 0 | 0 | 0 | 0
  Prothrombin Time, Grade 3 | 0 | 0 | 2 | 0
  Prothrombin Time, Grade 4 | 0 | 0 | 0 | 0
  Activated PartialThromboplastinTime(PTT) , Grade 1 | 3 | 0 | 10 | 1
  Activated PTT, Grade 2 | 0 | 0 | 0 | 0
  Activated PTT, Grade 3 | 0 | 0 | 0 | 0
  Activated PTT, Grade 4 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With at Least a 2-grade Worsening From Baseline in Hematological Toxicities
Description: The number of participants with at least a 2-grade worsening from Baseline in hematological toxicities were assessed. Clinical hematological parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable. Baseline is defined as the value of the variable measured at Day 0 prior to dosing.
Time Frame: From the day of the first dose of study agent (Day 0) until Day 56 (single-dose) or until Day 70 (double-dose)
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Placebo - Single-Dose | Placebo - Double-Dose | Raxibacumab - Single-Dose | Raxibacumab - Double-Dose
Number analyzed (Participants) | 74 | 6 | 217 | 23
Participants
  Leukocytosis, any >=2-grade worsening | 1 | 0 | 2 | 0
  Leukopenia, any >=2-grade worsening | 0 | 0 | 1 | 0
  Neutropenia, any >=2-grade worsening | 1 | 0 | 2 | 0
  Lymphopenia, any >=2-grade worsening | 0 | 0 | 1 | 0
  Hemoglobin, any >=2-grade worsening | 0 | 0 | 0 | 0
  Platelet, any >=2-grade worsening | 0 | 0 | 0 | 0
  Prothrombin Time, any >=2-grade worsening | 0 | 0 | 2 | 0
  Activated PTT, any >=2-grade worsening | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Liver Toxicities of the Indicated Grade
Description: Liver function parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable.
Time Frame: From the day of the first dose of study agent (Day 0) until Day 56 (single-dose) or until Day 70 (double-dose)
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Placebo - Single-Dose | Placebo - Double-Dose | Raxibacumab - Single-Dose | Raxibacumab - Double-Dose
Number analyzed (Participants) | 74 | 6 | 217 | 23
Participants
  Aspartate amino transferase (AST), Grade 1 | 2 | 0 | 7 | 0
  AST, Grade 2 | 0 | 0 | 0 | 0
  AST, Grade 3 | 0 | 0 | 0 | 0
  AST, Grade 4 | 0 | 0 | 0 | 0
  Alanine amino transferase(ALT), Grade 1 | 1 | 0 | 6 | 1
  ALT, Grade 2 | 0 | 0 | 0 | 0
  ALT, Grade 3 | 0 | 0 | 1 | 0
  ALT, Grade 4 | 0 | 0 | 0 | 0
  Gamma-glutamyl-transferase (GGT), Grade 1 | 0 | 0 | 3 | 1
  GGT, Grade 2 | 0 | 0 | 0 | 0
  GGT, Grade 3 | 0 | 0 | 0 | 0
  GGT, Grade 4 | 0 | 0 | 0 | 0
  Alkaline Phosphatase(ALP), Grade 1 | 0 | 0 | 0 | 0
  ALP, Grade 2 | 0 | 0 | 0 | 0
  ALP, Grade 3 | 0 | 0 | 0 | 0
  ALP, Grade 4 | 0 | 0 | 0 | 0
  Hyperbilirubinemia, Grade 1 | 3 | 0 | 5 | 1
  Hyperbilirubinemia, Grade 2 | 0 | 0 | 0 | 0
  Hyperbilirubinemia, Grade 3 | 0 | 0 | 0 | 0
  Hyperbilirubinemia, Grade 4 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With at Least a 2-grade Worsening From Baseline in Liver Toxicities
Description: The number of participants with at least a 2-grade worsening from Baseline in liver toxicities were assessed. Liver function parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable. Baseline is defined as the value of the variable measured at Day 0 prior to dosing.
Time Frame: From the day of the first dose of study agent (Day 0) until Day 56 (single-dose) or until Day 70 (double-dose)
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Placebo - Single-Dose | Placebo - Double-Dose | Raxibacumab - Single-Dose | Raxibacumab - Double-Dose
Number analyzed (Participants) | 74 | 6 | 217 | 23
Participants
  AST, any >=2-grade worsening | 0 | 0 | 0 | 0
  ALT, any >=2-grade worsening | 0 | 0 | 1 | 0
  GGT, any >=2-grade worsening | 0 | 0 | 0 | 0
  ALP, any >=2-grade worsening | 0 | 0 | 0 | 0
  Hyperbilirubinemia, any >=2-grade worsening | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Electrolyte Toxicities of the Indicated Grade
Description: Electrolyte function parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable.
Time Frame: From the day of the first dose of study agent (Day 0) until Day 56 (single-dose) or until Day 70 (double-dose)
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Placebo - Single-Dose | Placebo - Double-Dose | Raxibacumab - Single-Dose | Raxibacumab - Double-Dose
Number analyzed (Participants) | 74 | 6 | 217 | 23
Participants
  Hypernatremia, Grade 1 | 0 | 0 | 0 | 0
  Hypernatremia, Grade 2 | 0 | 0 | 0 | 0
  Hypernatremia, Grade 3 | 0 | 0 | 0 | 0
  Hypernatremia, Grade 4 | 0 | 0 | 0 | 0
  Hyponatremia, Grade 1 | 8 | 0 | 20 | 5
  Hyponatremia, Grade 2 | 0 | 0 | 0 | 0
  Hyponatremia, Grade 3 | 0 | 0 | 0 | 0
  Hyponatremia, Grade 4 | 0 | 0 | 0 | 0
  Hyperkalemia, Grade 1 | 3 | 0 | 3 | 3
  Hyperkalemia, Grade 2 | 0 | 0 | 0 | 0
  Hyperkalemia, Grade 3 | 0 | 0 | 0 | 0
  Hyperkalemia, Grade 4 | 0 | 0 | 0 | 0
  Hypokalemia, Grade 1 | 5 | 0 | 12 | 0
  Hypokalemia, Grade 2 | 0 | 0 | 0 | 0
  Hypokalemia, Grade 3 | 0 | 0 | 0 | 0
  Hypokalemia, Grade 4 | 0 | 0 | 0 | 0
  Hypomagnesemia, Grade 1 | 0 | 0 | 0 | 0
  Hypomagnesemia, Grade 2 | 0 | 0 | 0 | 0
  Hypomagnesemia, Grade 3 | 0 | 0 | 0 | 0
  Hypomagnesemia, Grade 4 | 0 | 0 | 0 | 0
  Hypercalcemia (HrC)/ adjusted for albumin, Grade 1 | 2 | 1 | 5 | 3
  HrC/ adjusted for albumin, Grade 2 | 0 | 0 | 1 | 0
  HrC/ adjusted for albumin, Grade 3 | 0 | 0 | 0 | 0
  HrC/ adjusted for albumin, Grade 4 | 0 | 0 | 0 | 0
  Hypocalcemia (HoC)/ adjusted for albumin, Grade 1 | 0 | 0 | 0 | 0
  HoC adjusted for albumin, Grade 2 | 0 | 0 | 0 | 0
  HoC/ adjusted for albumin, Grade 3 | 0 | 0 | 0 | 0
  HoC/ adjusted for albumin, Grade 4 | 0 | 0 | 0 | 0
  Hypercalcemia/ unadjusted, Grade 1 | 2 | 1 | 4 | 2
  Hypercalcemia/ unadjusted, Grade 2 | 0 | 0 | 1 | 0
  Hypercalcemia/ unadjusted, Grade 3 | 0 | 0 | 0 | 0
  Hypercalcemia/ unadjusted, Grade 4 | 0 | 0 | 0 | 0
  Hypocalcemia/ unadjusted, Grade 1 | 0 | 0 | 0 | 0
  Hypocalcemia/ unadjusted, Grade 2 | 0 | 0 | 0 | 0
  Hypocalcemia/ unadjusted, Grade 3 | 0 | 0 | 0 | 0
  Hypocalcemia/ unadjusted, Grade 4 | 0 | 0 | 0 | 0
  Hypophosphatemia, Grade 1 | 3 | 1 | 10 | 3
  Hypophosphatemia, Grade 2 | 1 | 0 | 5 | 0
  Hypophosphatemia, Grade 3 | 0 | 0 | 0 | 0
  Hypophosphatemia, Grade 4 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With at Least a 2-grade Worsening From Baseline in Electrolyte Toxicities
Description: The number of participants with at least a 2-grade worsening from Baseline in electrolyte toxicities were assessed. Electrolyte function parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable. Baseline is defined as the value of the variable measured at Day 0 prior to dosing.
Time Frame: From the day of the first dose of study agent (Day 0) until Day 56 (single-dose) or until Day 70 (double-dose)
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Placebo - Single-Dose | Placebo - Double-Dose | Raxibacumab - Single-Dose | Raxibacumab - Double-Dose
Number analyzed (Participants) | 74 | 6 | 217 | 23
Participants
  Hypernatremia, any >=2-grade worsening | 0 | 0 | 0 | 0
  Hyponatremia, any >=2-grade worsening | 0 | 0 | 0 | 0
  Hyperkalemia, any >=2-grade worsening | 0 | 0 | 0 | 0
  Hypokalemia, any >=2-grade worsening | 0 | 0 | 0 | 0
  Hypomagnesemia, any >=2-grade worsening | 0 | 0 | 0 | 0
  HrC/adjusted for albumin, any >=2-grade worsening | 0 | 0 | 1 | 0
  HoC/adjusted for albumin, any >=2-grade worsening | 0 | 0 | 0 | 0
  Hypercalcemia/unadjusted, any >=2-grade worsening | 0 | 0 | 1 | 0
  Hypocalcemia/unadjusted, any >=2-grade worsening | 0 | 0 | 0 | 0
  Hypophosphatemia, any >=2-grade worsening | 1 | 0 | 5 | 0

8. Primary Outcome: Number of Participants With Other Chemistry Toxicities of the Indicated Grade
Description: Other chemistry parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable.
Time Frame: From the day of the first dose of study agent (Day 0) until Day 56 (single-dose) or until Day 70 (double-dose)
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Placebo - Single-Dose | Placebo - Double-Dose | Raxibacumab - Single-Dose | Raxibacumab - Double-Dose
Number analyzed (Participants) | 74 | 6 | 217 | 23
Participants
  Creatinine, Grade 1 | 0 | 0 | 2 | 0
  Creatinine, Grade 2 | 0 | 0 | 0 | 0
  Creatinine, Grade 3 | 0 | 0 | 0 | 0
  Creatinine, Grade 4 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen (BUN), Grade 1 | 0 | 0 | 1 | 0
  BUN, Grade 2 | 0 | 0 | 0 | 0
  BUN, Grade 3 | 0 | 0 | 0 | 0
  BUN, Grade 4 | 0 | 0 | 0 | 0
  Hypoalbuminemia, Grade 1 | 3 | 0 | 1 | 0
  Hypoalbuminemia, Grade 2 | 0 | 0 | 0 | 0
  Hypoalbuminemia, Grade 3 | 0 | 0 | 0 | 0
  Hypoalbuminemia, Grade 4 | 0 | 0 | 0 | 0
  Hyperuricemia, Grade 1 | 1 | 0 | 8 | 0
  Hyperuricemia, Grade 2 | 0 | 0 | 1 | 0
  Hyperuricemia, Grade 3 | 0 | 0 | 0 | 0
  Hyperuricemia, Grade 4 | 0 | 0 | 0 | 0
  Hyperglycemia, Grade 1 | 15 | 0 | 36 | 8
  Hyperglycemia, Grade 2 | 1 | 0 | 1 | 2
  Hyperglycemia, Grade 3 | 0 | 0 | 0 | 0
  Hyperglycemia, Grade 4 | 0 | 0 | 0 | 0
  Hypoglycemia, Grade 1 | 5 | 0 | 11 | 2
  Hypoglycemia, Grade 2 | 2 | 0 | 2 | 3
  Hypoglycemia, Grade 3 | 0 | 0 | 0 | 0
  Hypoglycemia, Grade 4 | 0 | 0 | 0 | 0
  Amylase, Grade 1 | 5 | 0 | 25 | 2
  Amylase, Grade 2 | 4 | 0 | 5 | 1
  Amylase, Grade 3 | 0 | 0 | 1 | 0
  Amylase, Grade 4 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With at Least a 2-grade Worsening From Baseline in Other Chemistry Toxicities
Description: The number of participants with at least a 2-grade worsening from Baseline in other chemistry toxicities were assessed. Other clinical chemistry parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable. Baseline is defined as the value of the variable measured at Day 0 prior to dosing.
Time Frame: From the day of the first dose of study agent (Day 0) until Day 56 (single-dose) or until Day 70 (double-dose)
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Placebo - Single-Dose | Placebo - Double-Dose | Raxibacumab - Single-Dose | Raxibacumab - Double-Dose
Number analyzed (Participants) | 74 | 6 | 217 | 23
Participants
  Creatinine, any >=2-grade worsening | 0 | 0 | 0 | 0
  BUN, any >=2-grade worsening | 0 | 0 | 0 | 0
  Hypoalbuminemia, any >=2-grade worsening | 0 | 0 | 0 | 0
  Hyperuricemia, any >=2-grade worsening | 0 | 0 | 0 | 0
  Hyperglycemia, any >=2-grade worsening | 0 | 0 | 1 | 1
  Hypoglycemia, any >=2-grade worsening | 2 | 0 | 2 | 3
  Amylase, any >=2-grade worsening | 3 | 0 | 3 | 0

10. Primary Outcome: Number of Participants With Thyroid Toxicities of the Indicated Grade
Description: Clinical thyroid parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable.
Time Frame: From the day of the first dose of study agent (Day 0) until Day 56 (single-dose) or until Day 70 (double-dose)
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Placebo - Single-Dose | Placebo - Double-Dose | Raxibacumab - Single-Dose | Raxibacumab - Double-Dose
Number analyzed (Participants) | 74 | 6 | 217 | 23
Participants | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Participants With Urinalysis Toxicities of the Indicated Grade
Description: Urinaysis parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable.
Time Frame: From the day of the first dose of study agent (Day 0) until Day 56 (single-dose) or until Day 70 (double-dose)
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Placebo - Single-Dose | Placebo - Double-Dose | Raxibacumab - Single-Dose | Raxibacumab - Double-Dose
Number analyzed (Participants) | 74 | 6 | 217 | 23
Participants
  Proteinuria, Grade 1 | 9 | 0 | 31 | 3
  Proteinuria, Grade 2 | 3 | 0 | 9 | 0
  Proteinuria, Grade 3 | 0 | 0 | 0 | 0
  Proteinuria, Grade 4 | 0 | 0 | 0 | 0
  Hematuria, Grade 1 | 9 | 0 | 17 | 3
  Hematuria, Grade 2 | 4 | 0 | 15 | 2
  Hematuria, Grade 3 | 0 | 0 | 0 | 0
  Hematuria, Grade 4 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With at Least a 2-grade Worsening From Baseline in Urinalysis Toxicities
Description: Urinalysis parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable. Baseline is defined as the value of the variable measured at Day 0 prior to dosing.
Time Frame: From the day of the first dose of study agent (Day 0) until Day 56 (single-dose) or until Day 70 (double-dose)
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Placebo - Single-Dose | Placebo - Double-Dose | Raxibacumab - Single-Dose | Raxibacumab - Double-Dose
Number analyzed (Participants) | 74 | 6 | 217 | 23
Participants
  Proteinuria, any >=2-grade worsening | 3 | 0 | 8 | 0
  Hematuria, any >=2-grade worsening | 4 | 0 | 12 | 2

13. Primary Outcome: Number of Participants Who Developed an Anti-raxibacumab Antibody Response
Description: Number of participants who developed an anti-raxibacumab antibody response during the study were assessed. .Immunogenicity testing was performed to determine if raxibacumab induced an anti-raxibacumab immune response. Testing comprised of 2 assays (screening and confirmatory). The screening assay (direct binding) was an electrochemiluminescence (ECL)-based bridging assay. A rabbit polyclonal antibody was used as a positive control. Samples above the assay cut point were considered positive. Samples identified as positive in the screening assay were confirmed positive in a confirmatory assay. Samples must have demonstrated a significant percent drop in the confirmatory inhibition of binding assay to be considered positive. The inhibition of binding confirmatory assay was performed identically to the direct binding screening assay with the exception that the samples were tested in parallel with excess unlabeled raxibacumab.
Time Frame: From the day of the first dose of study agent (Day 0) until Day 56 (single-dose) or until Day 70 (double-dose)
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Placebo - Single-Dose | Placebo - Double-Dose | Raxibacumab - Single-Dose | Raxibacumab - Double-Dose
Number analyzed (Participants) | 74 | 6 | 217 | 23
Participants | 0 | 0 | 0 | 0

14. Secondary Outcome: Mean Raxibacumab Concentration-time Following a Single IV Infusion Dose
Description: Blood was collected from each participant at selected times post dose, and serum specimens were analyzed for raxibacumab using a validated electrochemiluminescense-based assay. The individual serum raxibacumab concentration data were summarized by nominal collection time and treatment group using descriptive statistics. Blood samples for serum raxibacumab concentration measurement were collected from participants who received a single-dose prior to administration of the raxibacumab and diphenhydramine doses on Day 0, at 30 minutes and 2 to 6 hours after completion of the raxibacumab infusion, and at 14, 28, and 56 days after the raxibacumab dose.
Time Frame: Pre-dose on Day 0, at 30 minutes and 2 to 6 hours after completion of raxibacumab infusion, and at 14, 28, and 56 days after the raxibacumab dose
Population: Pharmacokinetics (PK) Population: all evaluable participants who received a raxibacumab dose and had at least 1 measurable post-dose serum raxibacumab concentration.
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter (μg/mL)
Arm/Group | Raxibacumab - Single-Dose
Number analyzed (Participants) | 215
Micrograms per milliliter (μg/mL)
  Predose | 0.048 (0.631)
  30 minutes post-dose | 928.447 (191.293)
  2-6 hours post-dose | 881.586 (192.676)
  Day 14 | 311.669 (78.037)
  Day 28 | 199.043 (43.812)
  Day 56 | 89.021 (31.531)

15. Secondary Outcome: Mean Raxibacumab Concentration-time Following Two IV Infusion Doses
Description: Blood was collected from each participant at selected times post dose, and serum specimens were analyzed for raxibacumab using a validated electrochemiluminescense-based assay. The individual serum raxibacumab concentration data were summarized by nominal collection time and treatment group using descriptive statistics. For the participants that received two doses, blood samples for serum raxibacumab concentration measurement were collected from participants prior to administration of the raxibacumab and diphenhydramine doses on Days 0 and 14, at 30 minutes and 2 to 6 hours after completion of each raxibacumab infusion, and at 28, 42, 56, and 70 days after the 1st raxibacumab dose.
Time Frame: Pre-dose on Days 0 and 14, at 30 minutes and 2 to 6 hours after completion of each raxibacumab infusion, and at 28, 42, 56, and 70 days after the 1st raxibacumab dose
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter (μg/mL)
Arm/Group | Raxibacumab - Double-Dose
Number analyzed (Participants) | 23
Micrograms per milliliter (μg/mL)
  Dose 1 - Predose | 0 (0)
  Dose 1 - 30 minutes post-dose | 1012.564 (243.662)
  Dose 1 - 2-6 hours post-dose | 973.910 (261.825)
  Dose 2 - Predose | 314.374 (55.297)
  Dose 2 - 30 minutes post-dose | 1246.223 (224.481)
  Dose 2 - 2-6 hours post-dose | 1211.572 (210.793)
  Dose 2 - Day 14 | 543.767 (125.511)
  Dose 2 - Day 28 | 334.431 (78.980)
  Dose 2 - Day 42 | 213.463 (61.553)
  Dose 2 - Day 56 | 137.878 (46.231)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the time the first dose of study agent (Day 0) until Day 56 (single-dose) or until Day 70 (double-dose).
Description: SAEs and non-serious AEs were collected in the as-treated population, comprised of all participants randomized to treatment who received at least one dose of study agent.
Arm/Group | Placebo - Single-Dose | Placebo - Double-Dose | Raxibacumab - Single-Dose | Raxibacumab - Double-Dose
Serious Adverse Events (participants affected / at risk) | 0/74 | 1/6 | 0/217 | 1/23
Other Adverse Events (participants affected / at risk) | 32/74 | 6/6 | 103/217 | 10/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Single-Dose (N=74) | Placebo - Double-Dose (N=6) | Raxibacumab - Single-Dose (N=217) | Raxibacumab - Double-Dose (N=23)
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Single-Dose (N=74) | Placebo - Double-Dose (N=6) | Raxibacumab - Single-Dose (N=217) | Raxibacumab - Double-Dose (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Cardiac disorders (Cardiac disorders) | 0 | 1 | 2 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2 | 0
Blepharitis (Eye disorders) | 0 | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 4 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dental plaque (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 7 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Energy increased (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 3 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 1 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 1 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 1 | 0
Vessel puncture site paraesthesia (General disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 2 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 2 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 4 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 2 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 3 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 4 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 9 | 4
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Nerve injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood amylase increased (Investigations) | 0 | 0 | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 2 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 2 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 3 | 0
Headache (Nervous system disorders) | 7 | 1 | 19 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 2 | 1
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 2 | 0
Tension headache (Nervous system disorders) | 2 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Polymenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 5 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Hypertension (Vascular disorders) | 0 | 0 | 3 | 0
Pallor (Vascular disorders) | 1 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.